CLINICAL TRIAL: NCT06900153
Title: Description of Parental Projects, Pregnancies and Pregnancy Outcomes in Patients With a Classic Form of 21-hydroxylase Deficiency
Brief Title: Parenting and CAH - 21-hydroxylase Deficiency
Acronym: PARENT-HCS
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250491
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: CAH - 21-Hydroxylase Deficiency
Keywords: congenital adrenal hyperplasia due to 21; hydroxylase deficiency; fertility; pregnancy outcomes; pregnancy related; hormonal substitution; parental project
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: phone questionnaire — the investigator calls the patient and asks her questions about her parental project and her pregnancies

SUMMARY:
Congenital adrenal hyperplasia (CAH) is a genetic disease with autosomal recessive transmission, which is defined by a deficiency of one of the steroidogenesis enzymes. 21-hydroxylase deficiency (21OHD), related to mutations of the CYP21A2 gene, is involved in 90 to 95% of CAH cases. Depending on the severity of the mutations of this gene, there are severe forms known as "classic" (FC), with neonatal onset, and moderate forms known as "non-classic" (FNC), with onset later in childhood or after puberty. The classic form includes the salt-wasting form and the pure virilizing form, depending on the degree of aldosterone deficiency. The sexuality and fertility of women with classic 21OHD deficiency are impaired by several factors such as disruption of the gonadotropic axis due to overproduction of androgens and progesterone by the adrenal glands, and mechanical and psychological factors related to genital surgery. The fertility of these women improves over time, largely due to earlier treatment of CAH, improved therapeutic compliance and surgical advances in genital reconstruction leading to an increase in the percentage of patients who are sexually active. However, there is little data available, and even less on the course of pregnancy, its complications and its outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over
* Patients with HCS due to 21-hydroxylase deficiency, confirmed genetically
* Patients who have been informed and do not object to participating in the research

Exclusion Criteria:

* Patients who do not speak French
* Patients who are not affiliated to a social security scheme or who are not entitled to it
* Patients under legal protection, or under guardianship or trusteeship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with HCS due to 21-hydroxylase deficiency, confirmed genetically, and monitored in one of the participating Endocrinology departments affiliated with the CRMR of the FIRENDO network
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
to describe how pregnancies are achieved: spontaneous or induced, if induced by which ART technique. | Day 1
  Information on how the pregnancy was achieved will be collected from the medical file and will be supplemented on the day of inclusion by a telephone questionnaire to the patient

SECONDARY OUTCOMES:
Describe the existence of a parental project among the women in the cohort | Day 1
  The description of the parental project will be based on the patients' declaration of the presence or absence of a desire to have children, and if not, what the reasons were
Describe obstetric complications | Day 1
  The description of obstetrical complications (GEU, miscarriages, in utero fetal death, IUGR, gestational diabetes, hypertension, pre-eclampsia, HELLP syndrome, cholestasis gravidarum, term of delivery, spontaneous or induced labor, birth weight, breastfeeding if desired) will be based on data from pregnancy and childbirth follow-up reports.
Describe the hormonal substitution adjustments. | Day 1
  The description of hormone replacement adjustments will be based on the prescription of Hydrocortisone and Fludrocortisone.

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.